CLINICAL TRIAL: NCT04029779
Title: Evaluation of Immediately Placed Dental Implants With Local Application of Injectable-Platelet Rich Fibrin in Periodontally Compromised Sites. A Randomized Controlled Split Mouth Study
Brief Title: Evaluation of Immediately Placed Dental Implants With Local Application of Injectable PRF in Periodontally Compromised Sites
Acronym: PRF
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Krishnadevaraya College of Dental Sciences & Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 02_D012_81520
Record Dates: First submitted 2019-07-19; First posted 2019-07-23 (Actual); Last update posted 2019-12-12 (Actual); Status verified 2019-12

CONDITIONS: Bone Density; Bone Loss, Alveolar
Keywords: Injectable platelet rich fibrin; Bone density; Crestal bone loss; Immediate implants
MeSH Terms: conditions — Alveolar Bone Loss

STUDY DESIGN:
Intervention Model Description: Two groups were made one test and control. All the subjects were treated with immediate implants. In the test group subjects, injectable platelet-rich fibrin was coated around dental implants and was also injected in the socket. The control group received only dental implants.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Immediate implant placement coated with I-PRF (Experimental): The test group received implants coated with injectable platelet-rich fibrin and also the sockets were injected with injectable- platelet rich fibrin
  Interventions: Biological: I-PRF
- immediate implant only (No Intervention): The control group received immediate dental implants only after extraction of the teeth without any local coating.

INTERVENTIONS:
Biological: I-PRF — Local anaesthesia was administered and mucoperiosteal flap was reflected. Atraumatic tooth extraction was performed. Socket was curetted to remove the granulation tissue present in the socket with the help of curettes. The socket was well irrigated with saline. Implant osteotomies wasl performed with sequential drilling with standardized drills.I-PRF was freshly prepared 600rpm for 7 min(50g). 1ml of the i-PRF was applied in to the osteotomy site and the implant surface will be thoroughly coated followed by placing of the implant. The surgical site was thoroughly irrigated and debrided. Flap closure was achieved using 3-0 silk sutures to protect the implant site.
  Other Names: injectable platelet rich fibrin coated to dental implants.
  Arms: Immediate implant placement coated with I-PRF

SUMMARY:
The present study is a human, prospective, parallel, randomised controlled clinical trial conducted to explore the efficacy of injectable PRF around dental implants. The trial is in accordance with the Consolidated Standards of Reporting Trials (CONSORT) criteria, 2010.

DETAILED DESCRIPTION:
Ten healthy individuals satisfying the inclusion and exclusion criteria were recruited for the study. A detailed, thorough medical and dental history was obtained and each patient was subjected to comprehensive clinical and radiological examination. All patients were informed about the nature of the study, the surgical procedure involved, potential benefits and risks associated with the surgical procedure and written informed consent were obtained from all patients.

All the patients were treated with immediate implants. The injectable -PRF was coated on implants as well as injected in the socket in both the maxillary and mandibular anterior region. The clinical and radiographic parameters were recorded at baseline, three months and six months postoperatively.

ELIGIBILITY:
Inclusion Criteria:

1. Cooperative patients willing to participate in the study 2. At least two maxillary or mandibular anterior teeth indicated for extraction due to chronic periodontitis (chronic or aggressive) 3. Patients above 18 years of age 4. Patients with esthetic concerns 5. Patients with good oral hygiene maintenance 6. Adequate bone height apical to alveolus of the failing teeth (more than or equal to 5mm) to accommodate an implant

-

Exclusion Criteria:

1. Persistent & unresolved infection at implant site
2. Teeth with close proximity to anatomical structure and adjacent roots
3. Patients on radiotherapy
4. Patients with systemic disorders
5. Patients with parafunctional habits
6. Patients with history of alcohol, drug dependency and smoking

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2017-11-11 (Actual); Primary Completion 2019-11-30 (Actual); Study Completion 2019-11-30 (Actual)

PRIMARY OUTCOMES:
Crestal bone level | 6 months
  Measured using CBCT scan both on mesial and distal sides .The coronal surface of the implant will be taken as reference line from where two perpendicular lines are dropped on both mesial and distal aspect of implants to first bone to implant contact.
Bone density | 6 months
  measured using CBCT scan using Hounsfield units at mid point of the implant both on mesial and distal side with coronal portion of implant as reference line.

SECONDARY OUTCOMES:
Angular bleeding index | 6 months
  A periodontal probe passed along the buccal margin at 60 degrees angulation in gingival sulcus. The resultant bleeding is recorded as present (+) or absent (-).
Peri-implant Probing pocket depth | 6 months
  measured mesially and distally using a UNC-15 probe (university of North Carolina-15 periodontal probe- Hu-Friedy, Chicago, IL, USA).
Pink esthetic score | 6 months
  Digital photographs will be used for evaluation of the pink esthetic score(PES). Charts containing the seven variables will be designed. These include: mesial papilla, distal papilla, soft tissue level, soft tissue contour, alveolar process deficiency, soft tissue colour and texture. Each variable will be recorded with a 2-1-0 score, where 2 is the best and 0 is the poorest score.

CONTACTS AND LOCATIONS:
Locations (1):
- Krishnadevaraya college of dental sciences, Bangalore, Karnataka, India